CLINICAL TRIAL: NCT03264807
Title: A Multicenter Randomized Controlled Trial of D2 Versus D2 + Lymph Node 14v Dissection in Clinical Stage T3N+, T4N+ of Gastric Cancer (14VIGTORY Trial)
Brief Title: Lymph Node 14v Dissection in Clinical Stage T3N+, T4N+ of Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Hong Man Yoon, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015-0188
Record Dates: First submitted 2017-08-15; First posted 2017-08-29 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Gastric Cancer
Keywords: Lymph Node 14v; D2 lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 lymphadenectomy (Active Comparator): Subtotal gastrectomy with D2 lymphadnectomy (lymph node #1, #3, #4sb, #4d, #5, #6, #7, #8a, #9, #11p, #12a) could be performed in this arm
  Interventions: Procedure: D2 lymphadenectomy
- D2 and #14v lymphadenectomy (Experimental): Subtotal gastrectomy with D2 (lymph node #1, #3, #4sb, #4d, #5, #6, #7, #8a, #9, #11p, #12a) and lymph node #14v lymphadnectomy could be performed in this arm
  Interventions: Procedure: D2 and #14v lymphadenectomy

INTERVENTIONS:
Procedure: D2 lymphadenectomy — Subtotal gastrectomy with D2 lymphadenectomy (lymph node #1, #3, #4sb, #4d, #5, #6, #7, #8a, #9, #11p, #12a) is conventional surgery in patients with advanced gastric cancer such as T3N+ or T4N+ stage.
  Other Names: Subtotal gastrectomy
  Arms: D2 lymphadenectomy
Procedure: D2 and #14v lymphadenectomy — Subtotal gastrectomy with D2 (lymph node #1, #3, #4sb, #4d, #5, #6, #7, #8a, #9, #11p, #12a) and #14v lymphadenectomy is experimental surgery in patients with advanced gastric cancer such as T3N+ or T4N+ stage.
  Other Names: Subtotal gastrectomy; D2 lymphadenectomy; #14v lymphadenectomy
  Arms: D2 and #14v lymphadenectomy

SUMMARY:
The purpose of this study is to compare the survival rate according to the presence or absence of 14v lymph node dissection.

DETAILED DESCRIPTION:
The purpose of this study is to compare the survival rate according to the presence or absence of 14v lymph node dissection. Actually, if the 14v lymph node metastasis is suspected before surgery, it is excluded from the study. In a retrospective study conducted in our hospital, we compared the patients with the 14v lymphadenectomy group and those without the 14v lymphadenectomy group, the survival rate of the 14v lymphadenectomy group was 11% higher than that of the 14v non-lymphadenectomy group.Previous studies have suggested that the presence of metastatic lymph nodes in the 14v lymph node is not good and that removal of the 14v lymph node does not affect prognosis. However, if the lymph node is a continuous tissue and the transition to the 14v lymph node is confirmed microscopically, a negative prognosis may be expected because it is likely that the cancer has spread to the distal lymph node. In addition, inadequate resection of the lymphatic or 14v lymph node adjacent to the 14v lymph node in the absence of evidence of metastasis of the 14v lymph node under microscopic examination indicates that cancer may spread even after curative surgery, To prevent cancer metastasis.

ELIGIBILITY:
<Inclusion Criteria>

* Histologically proven primary gastric adenocarcinoma
* T3N+, T4N+ by CT scan (AJCC 7th classification)
* Distal margin of gastric cancer Location of distal margin of gastric cancer ; antrum, or angle of the stomach
* No evidence of other distant metastasis
* Age ≥ 20 year old
* Performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale
* No prior treatment of chemotherapy or radiation therapy against any other malignancies, and no prior treatment for gastric cancer including endoscopic mucosal resection
* Adequate organ functions defined as indicated below:

  1. WBC 3000/mm3 - 12,000/mm3
  2. > Serum Hemoglobin 8.0 g/dl
  3. > Serum Platelet 100 000/mm3
  4. < Serum AST 100 IU/l
  5. <Serum ALT 100 IU/l
  6. < Total Bilirubin 2.0 mg/dl
* Written signed informed consent

<Exclusion Criteria>

* Active double cancer (synchronous double cancer and metachronous double cancer within five disease-free years), excluding carcinoma in situ (lesions equal to intraepithelial or intramucosal cancer)
* Gastric remnant cancer
* Pregnant or breast-feeding women
* Mental disorder(diagnosed with mental disorder on medical record)
* Systemic administration of corticosteroids(include Herbal Medication)
* Unstable angina or myocardial infarction within 6 months of the trial
* Unstable hypertension
* Severe respiratory disease requiring continuous oxygen therapy
* Indications Total gastrectomy
* Borrmann type IV in the preoperative examination (including localized)
* Suspected LN # 14v metastasis during surgery
* Indications Pancreatectomy
* Suspected a metastasis of CT scans LN # 13, LN # 14
* Clinical stage IV group is suspected or confirmed during surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2015-08-06 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Superiority verification of disease-free survival after lymphadenectomy for D2 + 14v lymph node dissection in gastric resection in patients with T3N + and T4N + stomach cancer | the last recruited patient was followed up for 3 years
  Patients were randomized to an intention-to-treat population. The primary efficacy assessment was performed at the end of the 3-year follow-up period. The free-disease survival rates of the two groups were compared by log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: HONG MAN YOON, MD, Principal Investigator — National Cancer Center
Locations (12):
- South Korea (12):
  - The Catholic University of Korea, Incheon St. Mary'S Hospital, Incheon, Bupyeong-gu
  - Dongnam Inst. of Radiological & Medical Sciences, Busan, Gijang-gun
  - Gyeongsang national university hospital, Gyeongsang, Gingu-si
  - National Cancer Center, Gyeonggi-do, Goyang-si
  - catholic university of korea,Seoul ST. Mary's Hospital., Seocho, Seoul
  - Severance Hospital, Seoul, Sincon
  - Asan Medical Center, Seoul, Songpa-gu
  - A JOU University medical center, Gyeonggi-do, Suwon-si
  - Pusan National University Yangsan Hospital, Gyeongsang, Yangsan-si
  - Gyeongsang National University Changwon hospital, Changwon
  - Dankook University Hospital, Cheonan
  - The CATHOLIC University of KOREA, INCHEON ST.MARY's hospital, Incheon

IPD SHARING:
Plan to Share IPD: No